CLINICAL TRIAL: NCT01824316
Title: A Comparison of Management Strategies of Asthma in Pregnancy
Status: Completed | Type: Observational
Sponsor: Jennifer McCallister MD (Other)
Responsible Party: Sponsor-Investigator, Jennifer McCallister MD, Assistant Professor of Clinical Internal Medicine, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2012E0508
Record Dates: First submitted 2013-03-21; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Asthma; Pregnancy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Investigate differences in practice patterns in providers who may care for pregnant women with asthma exacerbations. The investigators believe that practitioners of different specialties will practice differently.

DETAILED DESCRIPTION:
The goal of this investigation is to determine how physicians manage pregnant patients with asthma exacerbations using patient vignettes. Vignettes or case studies have been shown in various areas of medicine to be an effective tool for surveying provider's knowledge and application of evidence-based guidelines (9,10,11,12). Specifically, we plan on surveying physicians-in-training and attending physicians in Emergency Medicine, Family Medicine, Internal Medicine, Obstetrics/Gynecology, and Pulmonary/Critical Care Medicine at the Ohio State University Werner Medical Center via electronic mail. Electronic mail addresses will be obtained from each Department or Division's Training Program Director. We have presented multiple, fictional, case-based scenarios and short, multiple-choice questions where the responder indicates how they would manage the case. No existing patient data will be used in the scenarios. In addition, demographic data of the physician including length of time in practice, numbers of patients seen with asthma exacerbations per month, and comfort level with the National Asthma Education and Prevention Program Guidelines (1). The survey is attached. Physicians who do not respond to the first electronic mail will be sent one follow-up electronic mail with a second request to complete the survey. Results from the questionnaires completed by each department/devision of physicians will be compared and analyzed for significant differences. The results will then be used to look for educational opportunities to improve the care of pregnant patients with asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Physicians-in-training and attending physicans at the Ohio State University Medical Center Emergency Medicine, Family Medicine, Internal Medicine, Obstetrics/Gynecology, and Pulmonary/Critical Care Medicine at the Ohio State University Werner Medical Center

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians-in-training and attending physicians in Emergency Medicine, Family Medicine, Internal Medicine, Obstetrics/Gynecology, and Pulmonary/Critical Care Medicine at the Ohio State University Werner Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Physician practice patterns in asthma management using clinical vignettes | Single use survey open for three month period
  The goal of this investigation is to determine how physicians manage pregnant patients with asthma exacerbations using patient vignettes. We have presented multiple, fictional, case-based scenarios and short, multiple-choice questions where the responder indicates how they would manage the case.

SECONDARY OUTCOMES:
Demographic description of respondents | Single use survey open for three month period
  Demographic data of physician respondents including length of time in practice, numbers of patients seen with asthma exacerbations per month, and comfort level with the National Asthma Education and Prevention Program Guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States